CLINICAL TRIAL: NCT01533454
Title: A Randomized Incentive-Based Weight Loss Trial in Singapore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0742_001
Record Dates: First submitted 2012-02-12; First posted 2012-02-15 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Incentives
Keywords: Obesity; Weight loss; Incentives; Motivation
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control participants will attend a 4-month structured weight-loss program and attend subsequent follow-ups at 4-month intervals upon completion of the program.
- Incentives (Experimental): Incentive arm participants will be offered an additional program (in addition to the COMM program) where they can earn incentives for meeting specified weight loss targets or step goals. They will be offered a choice between traditional (payments with certainty) and behavioral(payments paid via lottery) incentives.
  Interventions: Other: Financial Incentives

INTERVENTIONS:
Other: Financial Incentives — Incentive arm participants will be able to earn incentives for meeting specified weight loss targets or step goals. They will be offered a choice between traditional (payments with certainty) and behavioral(payments paid via lottery) incentives.
  Arms: Incentives

SUMMARY:
The purpose of this study is to test the extent to which incentives, when combined with an existing evidence-based weight loss program, improve weight loss and weight loss maintenance. It will also compare the cost-effectiveness of the incentive-based weight loss programs to the basic program without incentives.

DETAILED DESCRIPTION:
Globally, the rise in obesity rates has reached epidemic proportions, and in Singapore 53% of adults have a body mass index (BMI) great than 23.0 kg/m2, a level that increases risk for chronic disease among Asians. This study aims to test the extent to which traditional or behavioural economic incentives, when combined with an existing evidence-based weight loss program, improve weight loss and weight loss maintenance. Data will be collected through a two-arm (basic weight loss program, basic program plus traditional or behavioural economic incentives) randomized controlled trial (RCT) where key outcome variables are defined as weight loss (kilograms) at 8 months when the incentive program concludes, and at 12 months, after a 4 month period in which no additional incentives are provided. We hypothesize that at both 8 and 12 months, weight loss will be greater in the incentive arm than in the arm without incentives. The growing obesity epidemic, the high costs of obesity to employers, insurers and governments across Asia, and the fact that the incentive program is designed to be close to cost neutral, suggest that this research has high potential to have a significant public health impact, both in Singapore and the region.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 21+
* BMI 25+
* Willing to be randomized into 1 of the 2 study arms
* Willing to pay the $399 entry fee
* Stated willingness to commit to participating in all assessments regardless of weight change or study arm

Exclusion Criteria:

* Current pregnancy/lactation (women who become pregnant during the study will be withdrawn)
* Type 1 diabetes
* Type 2 diabetes on medication other than Metformin
* End-stage Renal Disease
* Ischemic Heart Disease requiring intervention in the past 6 months
* Thyroid disease that has yet to stabilize
* Changes in weight of greater than 3% in the past 6 months
* Use of weight loss medication in the past 6 months
* Malignancy requiring chemotherapy/radiation in the past 5 years
* Acute medical problems requiring 3+ days of missed work during previous 4 week period
* Any serious hospitalization or surgery in the past 6 months
* Use of corticosteroids in the past 6 months
* Answer 'YES' to any of the PAR-Q questions
* Unable to obtain MD consent from a physician giving permission to participate in the study
* Evidence of clinical depression (as assessed by the Beck Depression Inventory)
* Currently on medications for a mental health or substance abuse condition
* Evidence of binge eating based on the Binge Eating Disorders Scale (BEDS)
* Unable to communicate in English
* Additional concerns in which the clinical investigator deems problematic for participation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2012-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Weight change | Baseline, 4 months, 8 months and 12 months

SECONDARY OUTCOMES:
Percent body fat | Baseline, 4 months, 8 months, 12 months
Self-reported physical activity | Baseline, 4 months, 8 months, 12 months
Steps, aerobic steps and minutes of physical activity | Monthly through month 8 (in incentive arms)
Intrinsic and Extrinsic motivation | Baseline
Sociodemographics | Baseline
Health-related quality of life | Baseline, 4 months, 8 months, 12 months
Intervention costs | Baseline through month 8

CONTACTS AND LOCATIONS:
Overall Officials: Eric A. Finkelstein, PhD, MHA, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Finkelstein EA, Tham KW, Haaland BA, Sahasranaman A. Applying economic incentives to increase effectiveness of an outpatient weight loss program (TRIO) - A randomized controlled trial. Soc Sci Med. 2017 Jul;185:63-70. doi: 10.1016/j.socscimed.2017.05.030. Epub 2017 May 15. PMID 28554160